CLINICAL TRIAL: NCT00872651
Title: Travoprost 0.004%/Timolol 0.5% Versus Latanoprost 0.005%/Timolol in Chinese Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-08-074
Record Dates: First submitted 2009-02-25; First posted 2009-03-31 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; intraocular pressure; travoprost/timolol; timolol
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost 0.004%/Timolol 0.5% (Experimental): Travoprost 0.004%/Timolol 0.5%
  Interventions: Drug: Travoprost 0.004%/Timolol 0.5%
- Latanoprost 0.005% / Timolol 0.5% (Active Comparator): Latanoprost 0.005% / Timolol 0.5%
  Interventions: Drug: Latanoprost 0.005% / Timolol 0.5%

INTERVENTIONS:
Drug: Travoprost 0.004%/Timolol 0.5% — Travoprost 0.004%/Timolol 0.5%
  Arms: Travoprost 0.004%/Timolol 0.5%
Drug: Latanoprost 0.005% / Timolol 0.5% — Latanoprost 0.005% / Timolol 0.5%
  Arms: Latanoprost 0.005% / Timolol 0.5%

SUMMARY:
Eligible patients will be randomized in a 1.1 ratio to receive Travoprost 0.004%/timolol 0.5% once daily or Latanoprost 0.005%/Timolol 0.5% once a day for 8 Weeks. The study treatments will be compared for mean diurnal intraocular pressure (IOP) change from baseline at Week 8.

Safety parameters measured at 4 study visits: ocular signs, visual acuity, dilated fundus, cardiovascular parameters (blood pressure and pulse), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex and any race, 18 years of age or older, diagnosed with open angle glaucoma or ocular hypertension who are not sufficiently responsive to topical beta-blockers or prostaglandin analogues.
* Patients must meet the following IOP criteria in at least one eye. For each qualifying eye, the mean IOP should be ≥21 mmHg at 9 AM and 11 AM time points at the eligibility visit
* The mean IOP in either eye at the eligibility visit must not be greater than 35 mmHg at any time point.

Exclusion Criteria:

* Patients with any form of glaucoma other than open-angle glaucoma (with or without a pigment dispersion or pseudoexfoliation component) or ocular hypertension.
* Patients with iridocorneal angle Shaffer grade < 2 (extreme narrow angle with complete or partial closure) angle in either eye, as measured by gonioscopy
* Patients with a cup/disc ratio greater than 0.80 (horizontal or vertical measurement) in either eye.
* Patients with severe central visual field loss in either eye. Severe central field loss is defined as a sensitivity of ≤ 10 dB in at least 2 of the 4 visual field test points closest to the point of fixation.
* Current chronic, recurrent or severe inflammatory eye disease (e.g., scleritis, uveitis, herpes keratitis), or current other severe ocular pathology (including severe dry eye) that would affect the conduct of the study.
* History of ocular trauma within the past 6 months.
* Intraocular surgery within the past 3 months.
* Ocular laser surgery within the past 3 months.
* Best-corrected visual acuity score worse than 55 ETDRS letters read (equivalent to approximately 20/80 Snellen or 0.25 decimal)
* Current ocular infection or inflammation, or history of ocular infection or inflammation within the past 3 months, as determined by patients' history and/or examination.
* History of or current clinically relevant or progressive retinal disease, such as retinal degeneration, diabetic retinopathy or retinal detachment.
* Any abnormality preventing reliable applanation tonometry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 8 weeks
  Mean Diurnal Intraocular Pressure (IOP) (averaged at 9 AM, 11 AM and 4 PM) change from baseline at Week 8.

SECONDARY OUTCOMES:
Intraocular Pressure (IOP) | 8 weeks
  Mean IOP change from baseline at 9 AM at Week 2 and Week 6 visits and at 9 AM, 11 AM and 4 PM at Week 8 visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China